CLINICAL TRIAL: NCT00929045
Title: Growth Hormone and Insulin Growth Factor 1 Deficiencies in Children/Adolescents Following Traumatic Brain Injury: The Impact on Growth and Neuropsychological Recovery
Brief Title: Growth Hormone and Insulin Growth Factor 1 Deficiencies in Children/Adolescents Following Traumatic Brain Injury: The Impact on Growth and Neuropsychological Development
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Virginia Commonwealth University (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13239
Record Dates: First submitted 2009-06-24; First posted 2009-06-26 (Estimated); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Traumatic Brain Injury
Keywords: Growth Hormone replacement; subject 8 to 21; moderate to severe traumatic brain injury; growth hormone deficient
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Growth Hormone (Experimental)
  Interventions: Drug: Growth Hormone Replacement

INTERVENTIONS:
Drug: Growth Hormone Replacement

SUMMARY:
The purpose of this study is to look at the relationship between growth hormones, and recovery from a TBI - traumatic brain injury. It is believed that a TBI may interfere with the body's ability to produce growth hormones. These hormones may be needed by the body for growth, mental development and sexual maturation.

ELIGIBILITY:
Inclusion Criteria:

* This is Phase II trial-subjects have already completed Phase I.
* Traumatic brain injury (TBI).
* Results of the blood work from Phase I shows that your growth hormone levels are low.

Exclusion Criteria:

* Have not completed Phase I of the study.

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2007-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Neurocognitive changes following moderate/severe TBI | 1 year

IPD SHARING:
Plan to Share IPD: No